CLINICAL TRIAL: NCT03658369
Title: To Assess the Lanconone® (E-OA-07) Efficacy in Weight-bearing Joint Pain
Brief Title: Effect of LANCONONE in Weight-bearing Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EB/180601/LANCONONE/PAIN
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-09

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lanconone® (Active Comparator): Lanconone®: 2 Capsules once a day after breakfast
  Interventions: Dietary Supplement: Lanconone®
- Methyl Crystalline Cellulose (Placebo Comparator): 2 Capsules once a day after breakfast
  Interventions: Dietary Supplement: Methyl crystalline cellulose

INTERVENTIONS:
Dietary Supplement: Lanconone® — 2 capsules
  Arms: Lanconone®
Dietary Supplement: Methyl crystalline cellulose — 2 Capsules
  Arms: Methyl Crystalline Cellulose

SUMMARY:
The current study has been designed to primarily assess the effect of Lanconone® in comparison to placebo on pain in weight bearing joints.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 25 and ≤ 29.9 kg/m2.
2. With unilateral or bilateral OA of the knee for at least greater than 3 months, as presented by pain in the knee at least for last 3 months.
3. Post-menopausal females (LMP at least 12 months prior to the screening).

Exclusion Criteria:

1. History of osteoarthritis for more than 3 years.
2. Systolic Blood Pressure ≥140 mm Hg and Diastolic Blood Pressure ≥ 90 mm Hg
3. FBS>140 mg/dl.
4. Smokers or chronic alcoholics.
5. Participants planning to travel in the next 56 days or engage in any non-routine activity that is likely to strain the knees.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster universities Osteoarthritis Index) pain score | 56 days
  Change in pain score.The score ranges from 0-5, wherein 0 indicates no pain and 5 indicates extreme pain.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastava, M.D., Study Director — Vedic Lifesciences
Locations (4):
- India (4):
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Dinanath Nursing Home, Mumbai, Maharashtra
  - K.K Medical Centre, Mumbai, Maharashtra
  - Siddhant Clinic, Mumbai, Maharashtra